CLINICAL TRIAL: NCT04503772
Title: Phase II Study to Assess Preoperative Hypofractionated Stereotactic Radiotherapy of Brain Metastases
Brief Title: Preoperative Stereotactic Radiosurgery for Brain Metastases
Acronym: STEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Jean Perrin (Other)
Collaborators: Groupement Interrégional de Recherche Clinique et d'Innovation (AURA) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A00403-36; 20.06.16-36701 (Other: Ethics committee Sud-Ouest et Outre-Mer IV)
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Brain Metastases
Keywords: brain metastases; preoperative stereotactic radiosurgery; local control; radionecrosis; overall survival
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (all patients) (Experimental): Patients will receive preoperative hypofractionated stereotactic radiosurgery (SRS).
  According to the association of french-speaking neuro-oncologists (ANOCEF) recommendations, total dose and fractionation will be 33 Gy in 3 fractions at the isocenter, 23.1 Gy in envelope (70% isodose), i.e. 30 Gy in growth tumor volume (GTV) envelope.) Surgery will take place within 3 days of the preoperative SRS.
  Interventions: Procedure: Preoperative SRS

INTERVENTIONS:
Procedure: Preoperative SRS — Patient will be treat with preoperative SRS and then surgery for brain metastases is realized within 3 days.

SUMMARY:
STEP is a French multicentre, prospective, non-randomized, phase II study designed to assess 6-months local control after pre-operative stereotactic radiosurgery (SRS) for patients with brain metastases

ELIGIBILITY:
Inclusion Criteria:

* ≤ 4 distinct brain metastases, one with surgical indication
* Diagnosis of primary histologically proven breast, digestive or non-small cells lung cancer
* ≤ 5 cm larger diameter
* Karnofsky performance status ≥ 70
* No contraindication for MRI
* Possibility for the patient to be treat with both surgery and stereotactic radiotherapy
* ≥ 18 years old
* Estimated overall survival ≥ 6 months according to diagnosis specific - graded prognostic assessment (DS GPA)
* Written inform consent signed
* Affiliation to the French social security system
* For women of childbearing age including those on luteinizing hormone-releasing hormone (LH-RH) agonists for ovarian suppression: inclusion negative serum pregnancy test (≤ 7 days prior to the start of preoperative stereotactic radiosurgery (SRS).

Exclusion Criteria:

* Lymphoma, leukaemia, multiple myeloma, germinal tumours or cerebral primary cancer
* Metastases from small-cells lung cancer, kidney cancer, melanoma or sarcoma
* Mass effect with deflection ≥ 5 mm from median line or hydrocephaly or compression 4th ventricle, patient neurologically unstable, need for emergency decompressive surgery
* > 4 brain metastases
* Contraindication to anaesthesia, MRI or gadolinium injection
* Proximity of the tumour with organs at risk which do not allow the prescribed dose to be reached in the envelope
* Pregnant or breastfeeding woman
* Anti vascular endothelial growth factor (VEGF) within 6 weeks before treatment
* Documented leptomeningeal injury
* History of irradiation of the encephalon in toto
* History of stereotactic radiotherapy on metastasis to be operated on
* Non-candidate patient for surgery
* Surgical delay > 3 days compared to stereotactic radiotherapy
* Estimated survival < 6 months by DS GPA
* Patient under guardianship or curators
* Psychological disorder (cognitive disorders, mental alertness, etc.) or social (deprivation of liberty by judicial or administrative decision) or geographical reasons that may compromise medical monitoring of the trial or compliance with treatment
* Woman of childbearing age without effective contraception
* Patient participating in another intervention study within 4 weeks prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of 6-months local control rate after preoperative SRS | 6 months after preoperative SRS (M6)
  Local recurrence is defined as the onset or progression of nodular contrast grafting within the resection cavity according to the Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria.

SECONDARY OUTCOMES:
Evaluation of 1-year local control rate after preoperative SRS | 12 months after preoperative SRS (M12)
  Local recurrence is defined as the onset or progression of nodular contrast grafting within the resection cavity according to the RANO-BM criteria.
Evaluation of 1-year radionecrosis rate after preoperative SRS | 12 months after preoperative SRS (M12)
  Radionecrosis is defined either histologically post-operatively according to the anatomopathological report or in the absence of salvage surgery by the appearance or increase of gadolinium contrast on T1 MRI sequences associated with an increase in the cerebral brain volume (CBV) ratio (brain blood volume of the tumour / brain blood volume of the non-tumour white matter) of less than 2 on perfusion MRI sequences and/or a standard uptake volume (SUV max) of less than 1, 59 on positron emission tomography (PET) scanners at 6-fluoro-[18 fluoro]-L-dihydroxyphenylalanine (F-DOPA)
Evaluation of overall survival | At each follow-up visits after preoperative SRS : +3 months (M3); +6 months (M6); +9 months (M9); +12 months (M12)
  defined as the time interval between the date of preoperative radiosurgery and the date of death from any cause.
Evaluation of acute (less than 3 months post preoperative SRS) and delayed toxicities (more than 3 months after preoperative SRS) | At each follow-up visits after preoperative SRS : +3 months (M3); +6 months (M6); +9 months (M9); +12 months (M12)
  They will be collected and graded according to the NCI-CTCAE v5.0 scale. An adverse event of grade ≥ 3 will be considered "severe".
Rate of leptomeningeal relapses | At each follow-up visits after preoperative SRS : +3 months (M3); +6 months (M6); +9 months (M9); +12 months (M12)
  According to cerebral MRI
Evaluation of cerebral distant control | At each follow-up visits after preoperative SRS : +3 months (M3); +6 months (M6); +9 months (M9); +12 months (M12)
  Follow by MRI
Determination of predictive factors for local brain control, complication and prognosis factors for survival | At each follow-up visits after preoperative SRS : +3 months (M3); +6 months (M6); +9 months (M9); +12 months (M12)
Evaluation of cognitive function | At each follow-up visits after preoperative SRS : +3 months (M3); +6 months (M6); +9 months (M9); +12 months (M12)
  Mini-mental state examination (MMSE)
Evaluation of quality of life | At each follow-up visits after preoperative SRS : +3 months (M3); +6 months (M6); +9 months (M9); +12 months (M12)
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-Core 30 (C30)

CONTACTS AND LOCATIONS:
Overall Officials: Lucie BRUN, MD, Principal Investigator — Centre Jean Perrin
Locations (8):
- France (8):
  - Centre Jean PERRIN, Clermont-Ferrand, Puy-de-Dôme
  - CHU Grenoble Alpes, Grenoble
  - Hospices Civils de Lyon, Lyon
  - Centre Léon BÉRARD, Lyon
  - Centre Hospitalier d'Annecy-Genevois, Metz-Tessy
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Institut de cancérologie de la Loire Lucien Neuwirth, Saint-Priest-en-Jarez
  - Institut de cancérologie Strasbourg Europe (ICANS), Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ginzac A, Dupic G, Brun L, Molnar I, Casile M, Durando X, Verrelle P, Lemaire JJ, Khalil T, Biau J. Preoperative stereotactic radiosurgery for brain metastases: the STEP study protocol for a multicentre, prospective, phase-II trial. BMC Cancer. 2021 Jul 28;21(1):864. doi: 10.1186/s12885-021-08602-0. PMID 34320940
- See also: Study protocol article — https://pubmed.ncbi.nlm.nih.gov/34320940/